CLINICAL TRIAL: NCT03342001
Title: Assessing Quality of Life Changes Using Calcitonin in Patients With Hypothyroidism on Biochemical Replacement With Levothyroxine
Brief Title: Hypothyroidism Treated With Calcitonin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Kashif Munir, MD, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00076671
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Results first posted 2021-06-10 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Calcitonin; salmon calcitonin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment group, open label (Experimental): calcitonin nasal spray, 200 mcg daily
  Interventions: Drug: Calcitonin

INTERVENTIONS:
Drug: Calcitonin — calcitonin nasal spray
  Other Names: Miacalcin

SUMMARY:
Some people with hypothyroidism have persistent symptoms despite adequate treatment with thyroid hormones. We are testing whether giving calcitonin to such people will improve their quality of life.

DETAILED DESCRIPTION:
It is known that a proportion of patients with hypothyroidism despite serum TSH levels being within the normal reference range, may continue to express symptoms of hypothyroidism. Common symptoms include fatigue, muscle pain, weight gain, and mood changes. Saravanan et al. reported in a large community-based survey that patients on levothyroxine even with a normal TSH showed significant impairment in psychological well-being compared with age- and sex-matched controls. These patients are challenging to manage and are often unhappy with they care.

Established treatment of hypothyroidism is levothyroxine. Thyroid follicular cells synthesize and secrete thyroxine and triiodothyronine. However, even when people are receiving adequate levothyroxine replacement therapy, their quality of life may not improve. Calcitonin (CT) is also produced by the thyroid gland, parafollicular cells. Their levels are not tested in hypothyroidism because the exact role of calcitonin in human health and disease is not fully known. CT has long been thought to play an important role in bone and mineral homeostasis, particularly with respect to its ability to regulate calcium metabolism. CT has been found in fish, reptiles, birds, and mammals. Salmon-derived CT is 50-100 times more potent than human CT. Hence, salmon CT (sCT) has been used for medicinal purposes.

There is a need for further research in order to understand the nature of persisting symptoms in patients on T4 monotherapy despite a serum TSH within the reference range. Calcitonin has been shown to alleviate pain in patients with bone or mineral disorders. To date, the use of calcitonin for relief of hypothyroid symptoms has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Normal TSH on levothyroxine therapy

Exclusion Criteria:

1. pregnant or 6 months post partum
2. Current or previous thyroid cancer
3. Congenital hypothyroidism
4. any tobacco use
5. prescribed proton pump inhibitors
6. prescribed steroids
7. taking armour thyroid, naturethroid, or any dessicated thyroid hormone
8. Unstable medical conditions (CKD, Cirrhosis etc)
9. pituitary disease

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kashif Munir, M.D., Principal Investigator — University of Maryland
Locations (1):
- University of Maryland Center for Diabetes and Endocrinology, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saravanan P, Chau WF, Roberts N, Vedhara K, Greenwood R, Dayan CM. Psychological well-being in patients on 'adequate' doses of l-thyroxine: results of a large, controlled community-based questionnaire study. Clin Endocrinol (Oxf). 2002 Nov;57(5):577-85. doi: 10.1046/j.1365-2265.2002.01654.x. PMID 12390330

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group, Open Label
Started | 11
Completed | 9
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: people with hypothyroidism
Groups:
- Calcitonin: People with hypothyroidism
Arm/Group | Calcitonin
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Modified City of Hope Quality of Life Questionnaire for Patients With Thyroid Disease
Description: questionnaire to assess quality of life, 40 questions, 1-10 scale with 10 indicating more severe symptoms. Total 400 points, primary assessment was change in score after 6 weeks.
Time Frame: 6 weeks
Population: participants completing trial
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group, Open Label
Number analyzed (Participants) | 9
score on a scale | -36.33 (39.41)

ADVERSE EVENTS:
Time Frame: Only during trial 6 weeks per participant
Description: Low risk trial and no reasonable expectation of serious adverse event or mortality
Arm/Group | Treatment Group, Open Label
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group, Open Label (N=11)
nausea (Gastrointestinal disorders) | 1 (1)
kidney stone (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT03342001/Prot_SAP_000.pdf